CLINICAL TRIAL: NCT01181778
Title: Observational, Prospective, Multicenter Study to Evaluate the Educational Counseling Effects in the Choice of Different Combined Hormonal Contraceptives
Brief Title: Evaluation of Participant Responses to Educational Counseling About Different Combined Hormonal Contraceptive Choices (P06557)
Acronym: ECOS
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P06557
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2013-09-24 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Contraception
Keywords: hormonal contraceptive methods; combined hormonal contraceptive methods; physician counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Qualified Participants: All healthy women who consulted their physician for information on contraceptive choices and were eligible for primary and secondary outcome measure analysis, based on the physician's assessment

SUMMARY:
Physicians counsel women participants who are candidates for hormonal contraception about available combined hormonal contraceptive methods (the combined pill, the contraceptive vaginal ring [i.e., the etonogestrel + ethinylestradiol vaginal ring] and the contraceptive transdermal patch). Effects of this counseling on women's contraceptive use decisions are to be evaluated by 1) recording which method is chosen after information is provided about all three available combined hormonal methods, 2) comparing the final chosen contraceptive method used by a participant after counseling with the method originally intended to be used by that participant before the counseling, and 3) evaluating the criteria used by women participants to choose their contraceptive method after the counseling, including evaluation of social and demographic predictors of contraceptive choice. The differences among participants in the number of contacts made by the participants to physician offices for purposes of obtaining information regarding the use of their final chosen hormonal contraceptive (e.g., requests for clarification, questions, expressing doubt or reservations for using the method, or requests for other help/advisement by the physician) will also be evaluated over four months following the physician counseling.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women ≥ 18 years of age and ≤ 40 years of age who consult their physician for contraception and would consider a combined hormonal contraceptive method
* Women who are using the hormonal method for the first time or who have previously used and suspended it for at least 1 month
* Women on one combined pill who would consider switching to another combined pill (Women who attend their physician to stop one of the combined hormonal methods can not participate)
* Women who request a combined hormonal contraceptive method but for whom the physician considers another method more appropriate (e.g. contraindications for combined hormonal contraception) will be counseled about these methods but still complete the questionnaire
* Women who are not interested in becoming pregnant in the next 4 months
* Women who agree to complete a questionnaire and that the questionnaire data are reviewed and analyzed by staff participating in the project

Exclusion Criteria:

None

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women ≥ 18 years of age and < 40 years of age who consult their physician for information on contraception choices
Sampling Method: Non-Probability Sample
Enrollment: 1919 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

REFERENCES:
- [Result] Gambera A, Corda F, Papa R, Bastianelli C, Bucciantini S, Dessole S, Scagliola P, Bernardini N, de Feo D, Beligotti F. Observational, prospective, multicentre study to evaluate the effects of counselling on the choice of combined hormonal contraceptives in Italy--the ECOS (Educational COunselling effectS) study. BMC Womens Health. 2015 Sep 2;15:69. doi: 10.1186/s12905-015-0226-x. PMID 26329464

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants who were enrolled in the study
Period: Overall Study
Arm/Group | All Participants
Started | 1919
Completed | 1871
Not Completed | 48
Not completed — Physician Decision | 48

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 1919
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1919
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Choosing Each Hormonal Contraceptive Method Before and After Counseling
Description: Before receiving counseling, participants recorded on a questionnaire the method of contraception they thought they would choose. This was to be compared with the method of contraception the same participants thought they would choose after they received physician counseling, which was also recorded on their questionnaire.
Time Frame: Day of inclusion (Day 0) prior to physician counseling and after physician counseling
Population: The analysis population consisted of all participants who completed questionnaires before and after physician counseling and had no medical reason to prevent them from using a combined hormonal contraception method.
Measure: Number; unit: Participants
Groups:
- All Qualified Participants Before Counseling: Before counseling: All healthy women who were eligible for primary and secondary outcome measure analysis, based on the physician's assessment
- All Qualified Participants After Counseling: After counseling: All healthy women who were eligible for primary and secondary outcome measure analysis, based on the physician's assessment
Arm/Group | All Qualified Participants Before Counseling | All Qualified Participants After Counseling
Number analyzed (Participants) | 1871 | 1871
Participants
  Daily Pill | 1207 | 1199
  Weekly Patch | 60 | 131
  Monthy Ring | 97 | 397
  Other Method | 171 | 104
  Undecided | 336 | 40
Statistical Analysis 1: Comparison: All Qualified Participants Before Counseling vs All Qualified Participants After Counseling; Analysis of the difference in the percentage of participants who chose the Daily Pill before physician counseling and after physician counseling; Test type: Superiority or Other; p = 0.705, Chi-squared; Difference in Percentage: Daily Pill = -0.4, 95% CI 2-sided [-2.6 to 1.8]
Statistical Analysis 2: Comparison: All Qualified Participants Before Counseling vs All Qualified Participants After Counseling; Analysis of the difference in the percentage of participants who chose the Weekly Patch before physician counseling and after physician counseling; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference in Percentage: Weekly Patch = 3.8, 95% CI 2-sided [2.6 to 5.0]
Statistical Analysis 3: Comparison: All Qualified Participants Before Counseling vs All Qualified Participants After Counseling; Analysis of the difference in the percentage of participants who chose the Monthly Ring before physician counseling and after physician counseling; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference in Percentage: Monthy Ring = 16.0, 95% CI 2-sided [14.3 to 17.8]
Statistical Analysis 4: Comparison: All Qualified Participants Before Counseling vs All Qualified Participants After Counseling; Analysis of the difference in the percentage of participants who chose Other Method before physician counseling and after physician counseling; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference in Percentage: Other Method = -3.6, 95% CI 2-sided [-5.0 to -2.2]
Statistical Analysis 5: Comparison: All Qualified Participants Before Counseling vs All Qualified Participants After Counseling; Analysis of the difference in the percentage of participants who chose Undecided before physician counseling and after physician counseling; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference in Percentage: Undecided = -15.8, 95% CI 2-sided [-17.6 to -14.1]

2. Secondary Outcome: Percentage of Participants With Post-counseling Contacts With Physician Offices, by Hormonal Contraceptive Method
Description: Participant contacts with physician offices were collected, and the number of callbacks by method of contraception recorded. Participants who called back more than once were counted overall and for each method of contraception.
Time Frame: Up to four months after the counseling visit
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | All Qualified Participants
Number analyzed (Participants) | 1871
percentage of participants
  Daily Pill (n=1199) | 5.1
  Weekly Patch (n=131) | 6.9
  Monthly Ring (n=397) | 6.0
  Other Method (n=104) | 1.9
  Undecided (n=40) | 2.5

ADVERSE EVENTS:
Time Frame: Four months
Description: Of the 1919 participants enrolled in the study, 48 participants did not meet eligibility requirements for primary and secondary outcome measure analysis and safety analysis, based on physicians' assessments.
Groups:
- All Qualified Participants: All healthy women who consulted their physician for information on contraceptive choices and were eligible for primary and secondary outcome measure analysis and safety analysis, based on the physician's assessment
Arm/Group | All Qualified Participants
Serious Adverse Events (participants affected / at risk) | 0/1871
Other Adverse Events (participants affected / at risk) | 0/1871

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators have accepted and committed not to disclose

information herein contained. Investigators will not to publish or disclose any results pertaining to the study without written authorization by the Sponsor.

Investigators accept that the Sponsor will review any manuscript or abstract 30 days before submission for a publication or presentation (including oral

presentations) containing data derived from the present study.